CLINICAL TRIAL: NCT00519285
Title: A Multicenter, Randomized, Double Blind Study Comparing the Efficacy and Safety of Aflibercept Versus Placebo Administered Every 3 Weeks in Patients Treated With Docetaxel/ Prednisone for Metastatic Androgen-independent Prostate Cancer
Brief Title: Aflibercept in Combination With Docetaxel in Metastatic Androgen Independent Prostate Cancer
Acronym: VENICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC6546; 2006-004756-20 (EudraCT Number)
Record Dates: First submitted 2007-08-21; First posted 2007-08-22 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Prostatic Neoplasms; Neoplasm Metastasis
Keywords: metastatic; prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — aflibercept; Docetaxel; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo added to standard chemotherapy with docetaxel plus prednisone or prednisolone
  Interventions: Drug: Placebo (for aflibercept); Drug: Docetaxel; Drug: Prednisone or Prednisolone
- Aflibercept (Experimental): Aflibercept added to standard chemotherapy with docetaxel plus prednisone or prednisolone
  Interventions: Drug: Aflibercept; Drug: Docetaxel; Drug: Prednisone or Prednisolone

INTERVENTIONS:
Drug: Aflibercept — 25 mg/ml solution
  6 mg/kg, 1-hour IV on Day 1 of each 3-Week cycle
  Other Names: AVE0005; ZALTRAP®)
  Arms: Aflibercept
Drug: Placebo (for aflibercept) — Sterile aqueous buffered solution identical to aflibercept
  1-hour IV on Day 1 of each 3-Week cycle
  Arms: Placebo
Drug: Docetaxel — Marketed formulation
  75 mg/m², 1 hour IV on Day 1 of each 3-week cycle (immediately after Aflibercept or placebo)
  Other Names: Taxotere®
Drug: Prednisone or Prednisolone — Marketed formulation
  5 mg twice daily PO from day 1 continuously

SUMMARY:
Primary objective was to demonstrate overall survival improvement with aflibercept compared to placebo in patients receiving docetaxel / prednisone for metastatic androgen-independent prostate cancer (MAIPC).

The secondary objectives were:

* To assess the efficacy of aflibercept compared to placebo on other parameters such prostate-specific antigen (PSA) level, cancer related pain, progression free survival (PFS), tumor-based and skeletal events and health-related quality of life (HRQL);
* To assess the overall safety in both treatment arms;
* To determine the pharmacokinetics of intravenous (IV) aflibercept in this population;
* to determine immunogenicity of IV aflibercept.

DETAILED DESCRIPTION:
The study consisted in 3-week treatment cycles until progressive disease, unacceptable toxicity, or participant's refusal of further study treatment. After disease progression, participants were to be followed every 3 months until death or the study cutoff date, whichever came first.

The study cut-off date was event-driven and was defined as the date when 873 deaths had occurred.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed prostate adenocarcinoma;
* Metastatic disease;
* Progressive disease while receiving hormonal therapy or after surgical castration;
* Effective castration.

Exclusion Criteria:

* Prior cytotoxic chemotherapy for prostate cancer, except estramustine and except adjuvant/neoadjuvant treatment completed >3 years ago;
* Prior treatment with Vascular Endothelial Growth Factor (VEGF) inhibitors or VEGF receptor inhibitors;
* Eastern Cooperative Oncology Group (ECOG) performance status >2.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2007-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (31):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Providencia Santiago, Chile
- Sanofi-Aventis Administrative Office, City of Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Tallinn, Estonia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Gauteng, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Tannock IF, Fizazi K, Ivanov S, Karlsson CT, Flechon A, Skoneczna I, Orlandi F, Gravis G, Matveev V, Bavbek S, Gil T, Viana L, Aren O, Karyakin O, Elliott T, Birtle A, Magherini E, Hatteville L, Petrylak D, Tombal B, Rosenthal M; VENICE investigators. Aflibercept versus placebo in combination with docetaxel and prednisone for treatment of men with metastatic castration-resistant prostate cancer (VENICE): a phase 3, double-blind randomised trial. Lancet Oncol. 2013 Jul;14(8):760-8. doi: 10.1016/S1470-2045(13)70184-0. Epub 2013 Jun 4. PMID 23742877
- [Derived] van Soest RJ, Templeton AJ, Vera-Badillo FE, Mercier F, Sonpavde G, Amir E, Tombal B, Rosenthal M, Eisenberger MA, Tannock IF, de Wit R. Neutrophil-to-lymphocyte ratio as a prognostic biomarker for men with metastatic castration-resistant prostate cancer receiving first-line chemotherapy: data from two randomized phase III trials. Ann Oncol. 2015 Apr;26(4):743-749. doi: 10.1093/annonc/mdu569. Epub 2014 Dec 15. PMID 25515657
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2007 and February 2010, a total of 1548 patients gave informed consent for this study.
Pre-assignment Details: Amongst these patients, a total of 324 were screening failures (primarily due to non-compliance with exclusion criteria) and did not get randomized.
Groups:
- Placebo: Placebo, 1 hour IV, immediately followed by docetaxel, 75 mg/m² 1 hour IV, every 3 weeks in combination with oral prednisone or prednisolone, 5 mg PO twice daily
- Aflibercept: Aflibercept, 6 mg/kg 1 hour IV, immediately followed by docetaxel, 75 mg/m² 1 hour IV, every 3 weeks in combination with oral prednisone or prednisolone, 5 mg PO twice daily
Period: Overall Study
Arm/Group | Placebo | Aflibercept
Started | 612 (Randomized) | 612 (Randomized)
TREATED | 604 (Received at least part of one dose of placebo) | 605 (Received at least part of one dose of aflibercept)
Still Treated at Cut-off Date | 1 (The cut-off date for analysis was defined as 07 February 2012, date at which 873 deaths has occurred) | 2
Completed | 0 (Participants were treated until progressive disease, unacceptable toxicity, or refusal of treatment) | 0
Not Completed | 612 | 612
Not completed — Adverse Event | 127 | 266
Not completed — Disease progression | 334 | 186
Not completed — Physician Decision | 75 | 47
Not completed — Participant's request | 53 | 84
Not completed — Consent withdrawn | 4 | 5
Not completed — Poor compliance to protocol | 5 | 7
Not completed — Reason unspecified | 5 | 8
Not completed — Not treated | 8 | 7
Not completed — Treatment ongoing | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aflibercept | Total
Number analyzed (Participants) | 612 | 612 | 1224
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (8.0) | 67.9 (7.8) | 67.8 (7.9)
Age, Customized [Number; unit: participants]
  <65 years | 225 | 195 | 420
  65-74 years | 259 | 283 | 542
  ≥75 years | 128 | 134 | 262
Sex/Gender, Customized [Number; unit: participants]
  Male | 612 | 612 | 1224
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 552 | 560 | 1112
  Black | 17 | 15 | 32
  Asian/Oriental | 36 | 32 | 68
  Other | 7 | 5 | 12
Region of Enrollment [Number; unit: Participants]
  Western Europe | 219 | 227 | 446
  Eastern Europe | 131 | 132 | 263
  North America | 81 | 95 | 176
  South America | 88 | 71 | 159
  Other region | 93 | 87 | 180
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 2.0 (0.2) | 2.0 (0.2) | 2.0 (0.2)
Eastern Co-operative Group (ECOG) performance status [Number; unit: participants] — ECOG performance status:
  * 0 = Fully active, able to carry on all pre-disease performance without restriction
  * 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    ECOG 0 | 285 | 283 | 568
    ECOG 1 | 299 | 303 | 602
    ECOG 2 | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time
Description: Overall survival (OS) time was measured as the time from date of randomization to the date of death due to any cause.
  The median OS time and its 95.6% confidence interval were estimated using the Kaplan-Meier method. In the absence of confirmation of death, the participant was censored at the last date he/she was known to be alive or the study cut-off date (when 873 deaths have occurred), whichever was earlier.
Time Frame: From randomization up to the cut-off date (median follow-up of 35.4 months)
Population: The analysis was performed on the Intent-to-treat (ITT) population (i.e all randomized participants according to the treatment assigned regardless of the drug actually received).
  At the cut-off date, 873 deaths had occurred, 445 in the Placebo group and 428 in the Aflibercept group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 612 | 612
months | 21.22 [19.614 to 23.754] | 22.14 [20.304 to 24.082]
Statistical Analysis 1: Comparison: Placebo vs Aflibercept; Null hypothesis: No difference between aflibercept and placebo The study was designed to provide 90% power to detect a 1.25-fold increase in median survival with aflibercept compared to placebo at a overall one-sided significance level of 0.025 with 873 deaths; Test type: Superiority or Other; p = 0.3802, Log Rank — A priori threshold for statistical significance was set to 0.044 using the O'Brien-Fleming alpha spending function to account for two interim analyses; Log rank test stratified on ECOG Performance Status; Hazard Ratio (HR) = 0.942, 95.6% CI 2-sided [0.822 to 1.08] — Hazard ratio (HR) aflibercept versus placebo estimated from a Cox proportional hazard model stratified on ECOG Performance Status

2. Secondary Outcome: Prostate Specific Antigen Response Rate
Description: Prostate specific antigen (PSA) response was defined as ≥50% decrease from baseline in serum PSA levels, confirmed at least 3 weeks later. Increases of any magnitude during the first 12 weeks were ignored in determining PSA response.
Time Frame: Before randomization (baseline) then every 3 weeks up to PSA progression (≥25% increase) or the cut-off date, whichever occurred first
Population: The analysis was performed on the ITT population evaluable for PSA response (i.e. with a baseline PSA ≥10 ng/mL).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 559 | 560
percentage of participants | 63.5 [59.5 to 67.5] | 68.6 [64.7 to 72.4]

3. Secondary Outcome: Time to Skeletal Related Events
Description: Skeletal Related Events (SRE) included pathological fractures and/or spinal cord compression, need for bone irradiation, including radioisotopes or bone surgery, change in antineoplastic therapy to treat bone pain.
  Time to SRE was defined as the time from the date of randomization to the date of occurence of the first event defining a SRE or death due to any cause, whichever occurred first.
  The median time to SRE and its 95% confidence interval were estimated using the Kaplan-Meier method. In the absence of SRE, the participant was censored at the last date he/she was known to be alive or the study cut-off date, whichever was earlier.
Time Frame: From randomization up to the cut-off date (median follow-up of 35.4 months)
Population: The analysis was performed on the ITT population.
  At the cut-off date, SRE or death had occurred in 1013 participants, 516 in the Placebo group and 497 in the Aflibercept group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 612 | 612
months | 14.98 [13.733 to 16.427] | 15.31 [14.127 to 16.657]

4. Secondary Outcome: Progression Free Survival Time
Description: Disease progression was defined as a composite of: Radiological tumor progression (≥20% increase in target lesions, or appearance of at least 2 new bone lesions); PSA progression (≥25% increase in PSA level confirmed 3 weeks later); Pain progression (increase in pain intensity or in analgesic consumption for cancer related pain confirmed 3 weeks later); Radiotherapy for cancer related symptoms; Occurence of Skeletal related events (SRE).
  Progression Free survival (PFS) time was measured as the time from the date of randomization up to the date of occurrence of the first event defining a disease progression or death due to any cause, whichever occurred first.
  The median PFS time and its 95% confidence interval were estimated using the Kaplan-Meier method. In the absence of disease progression, the participant was censored at the the date of last assessment without evidence of progression or the study cut-off date, whichever was earlier.
Time Frame: From randomization up to the cut-off date (median follow-up of 35.4 months)
Population: The analysis was performed on the ITT population.
  At the cut-off date, disease progression or death had occurred in 1184 participants, 592 in each treatment group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 612 | 612
months | 6.24 [5.585 to 6.899] | 6.90 [6.209 to 7.359]

5. Secondary Outcome: Tumor Response Rate in Participants With Measurable Disease
Description: Tumor response was defined as either a Complete Response (disappearance of all target lesions) or a Partial Response (≥30% decrease from baseline in target lesions) as assessed by Response Evaluation Criteria In Solid Tumors (RECIST)version 1.0.
Time Frame: Before randomization (baseline) then every 3 months up to tumor progression (≥25% increase) or the cut-off date, whichever occurred first
Population: The analysis was performed on the ITT population evaluable for tumor response (i.e. received at least one dose of study drugs (aflibercept/placebo or docetaxel), had no important deviations to protocol and was evaluable for response as per RECIST version 1.0).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 320 | 323
percentage of participants | 28.1 [23.2 to 33.1] | 38.7 [33.4 to 44.0]

6. Secondary Outcome: Prostate Specific Antigen Progression-free Survival Time
Description: Prostate specific antigen (PSA) progression was defined as ≥25% increase in PSA level confirmed 3 weeks later, above the nadir in participants who had achieved a PSA response, or above the baseline in participants who hadn't achieved a PSA response.
  PSA progression-free survival (PFS) time was defined as the time from the date of randomization up to the date of the first documented PSA progression or death due to any cause, whichever occurred first.
  The median PSA-PFS time and its 95% confidence interval were estimated using the Kaplan-Meier method. In the absence of PSA progression or death, the participant was censored at the the date of last assessment without evidence of progression or the study cut-off date, whichever was earlier.
Time Frame: From randomization up to the cut-off date (median follow-up of 35.4 months)
Population: The analysis was performed in the ITT population evaluable for PSA progression (i.e. with an evaluable baseline PSA).
  At the cut-off date, PSA progression or death had occurred in 1138 participants, 571 in the Placebo group and 567 in the Aflibercept group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 606 | 608
months | 8.11 [7.622 to 8.575] | 8.25 [7.819 to 8.772]

7. Secondary Outcome: Pain Progression-free Survival Time
Description: Pain progression was defined as either ≥1-point increase in Present Pain Intensity (PPI) score or ≥25% increase in Analgesics Score (AS) confirmed at least 3 weeks later, or requirement for palliative radiotherapy. PPI scale is a self-report 0-5 scale to assess pain intensity - a score 0 reflects no pain, a score 5 reflects excruciating pain. AS is a scoring method to assess analgesics consumption. Each analgesic is scored 1 or 4 depending on the analgesic type and dose. AS is the sum of the analgesic scores.
  Pain progression-free survival (PFS) time was measured as the time from the date of randomization up to the date of first pain progression or death due to any cause, whichever occurred first.
  The median pain-PFS and its 95% confidence interval were estimated using the Kaplan-Meier method. In the absence of event, the participant was censored at the the date of last assessment without evidence of pain progression or the study cut-off date, whichever was earlier.
Time Frame: From randomization up to the cut-off date (median follow-up of 35.4 months)
Population: The analysis was performed on the ITT population evaluable for pain progression (i.e. with no pain or with stable pain at baseline).
  At the cut-off date, pain progression or death had occurred in 507 participants, 263 in the Placebo group and 244 in the Aflibercept group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 301 | 287
months | 9.72 [8.509 to 11.499] | 9.20 [8.181 to 10.448]

8. Secondary Outcome: Pain Response Rate
Description: Pain response was defined as either a ≥2-point decrease from baseline in Present Pain Intensity (PPI) score without increase in Analgesics Score (AS), or a ≥50% decrease from baseline in AS without increase in the PPI score confirmed at least 3 weeks later. Increases in PPI or AS during the first 12 weeks were ignored in determining pain response.
Time Frame: Before randomization (baseline) then every 3 weeks up to pain progression or the cut-off date, whichever occurred first
Population: The analysis was performed in the ITT population evaluable for pain response (i.e. stable analgesia at baseline and, baseline PPI ≥2 and/or baseline AS ≥10 points).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 67 | 67
percentage of participants | 46.3 [34.3 to 58.2] | 35.8 [24.3 to 47.3]

9. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate Total Score as a Measure of Health Related Quality of Life
Description: Functional Assessment of Cancer Therapy-Prostate (FACT-P) is a 39-item participant questionnaire that measures the concerns of patients with prostate cancer. It consists of 5 subscales assessing physical well-being, social/family well-being, emotional well-being, functional well-being, and prostate-specific concerns.
  FACT-P total score is the sum of the 5 subscores. It ranges from 0 to 156 with higher score indicating better quality of life.
Time Frame: Before randomization (baseline) then every 3 weeks until disease progression or administration of further antitumor therapy, whichever came first
Population: The analysis was performed on the ITT population evaluable for Health related quality of life (i.e. with baseline and at least one post-baseline evaluable FACT-P questionnaire).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 574 | 568
units on a scale
  Change from baseline at cycle 1 (n =493, 461) | 5.08 (12.73) | 1.30 (15.70)
  Change from baseline at cycle 2 (n =467, 437) | 6.22 (14.50) | -0.03 (17.99)
  Change from baseline at cycle 6 (n =293, 224) | 5.50 (16.38) | -1.00 (16.85)
  Change from baseline at cycle 10 (n =158, 117) | 6.61 (16.35) | -1.60 (15.41)

10. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Adverse Events (AE) are any unfavorable and unintended sign, symptom, syndrome or illness observed by the investigator or reported by the participant during the study.
  AE were collected at regular intervals throughout the study then graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v.3.0).
Time Frame: From first dose of study treatment (aflibercept/placebo or docetaxel whichever came first) to last dose of study treatment (aflibercept/placebo or docetaxel whichever came last) + 30 days
Population: The analysis was performed on the safety population (i.e. all randomized and treated participants according to the treatment actually received). Six participants in the Placebo group who received at least one dose of aflibercept in error were considered in the Aflibercept group.
Measure: Number; unit: participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 598 | 611
participants
  Any Adverse Event | 585 | 607
  - Grade 3-4 AE | 290 | 470
  - Serious AE | 184 | 331
  - AE leading to death | 23 | 46
  --- Related AE leading to death | 8 | 19
  - AE leading to permanent discontinuation | 125 | 268
  - AE leading to premature discontinuation | 73 | 116

11. Secondary Outcome: Number of Participants With Positive Anti-aflibercept Antibody Levels as a Measure of Immunogenicity of Aflibercept
Description: Serum for detection of anti-drug antibodies (ADA) was collected in patients treated in selected centers only. Samples were analyzed using a titer-based, bridging immunoassay developed and validated to detect ADAs in human serum.
  Samples with positive antibody levels were further analyzed using a validated, non-quantitative ligand binding assay to detect neutralizing antibodies Ab).
  A participant was considered to have positive antibody levels if antibodies were detected above the quantification limits.
Time Frame: Pre-dose of cycle 1 (baseline), pre-dose of each every other cycle, then 30 and 90 days after the last administration of the study drug
Population: The analysis was performed on the safety population evaluable for immunogenicity (i.e. exposed to aflibercept with serum samples evaluable for immunogenicity).
Measure: Number; unit: participants
Arm/Group | Placebo | Aflibercept
Number analyzed (Participants) | 149 | 179
participants
  At baseline | 0 | 2
  At any time post-baseline | 4 | 9
  - Neutralizing Ab | 0 | 2
  - Not neutralizing Ab | 2 | 5
  - Neutralizing potential not evaluated | 2 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected from signature of the informed consent form up to the last visit in the study.
Description: The analysis was performed on the safety population as described for Outcome measure 10 (i.e. according to the treatment actually received) and included all AE that developed or worsened from first dose of aflibercept/placebo or docetaxel whichever came first, to 30 days after last dose of aflibercept/placebo or docetaxel whichever came last.
Arm/Group | Placebo | Aflibercept
Serious Adverse Events (participants affected / at risk) | 184/598 | 331/611
Other Adverse Events (participants affected / at risk) | 551/598 | 573/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=598) | Aflibercept (N=611)
Urinary tract infection (Infections and infestations) | 4 | 10
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 11 | 21
Neutropenic infection (Infections and infestations) | 12 | 22
Bronchitis (Infections and infestations) | 1 | 2
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 13
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Localised infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 3 | 7
Sepsis (Infections and infestations) | 2 | 4
Gastroenteritis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 4
Skin infection (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 3
Device related infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 2
Peridiverticular abscess (Infections and infestations) | 0 | 3
Rectal abscess (Infections and infestations) | 0 | 3
Abscess intestinal (Infections and infestations) | 0 | 2
Abscess limb (Infections and infestations) | 1 | 0
Anal infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 2
Abdominal abscess (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Nasal abscess (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyonephrosis (Infections and infestations) | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0
Cystitis bacterial (Infections and infestations) | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0
Herpes oesophagitis (Infections and infestations) | 0 | 1
Infected bites (Infections and infestations) | 0 | 1
Infectious peritonitis (Infections and infestations) | 0 | 1
Listeria sepsis (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
West nile viral infection (Infections and infestations) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 21 | 48
Neutropenia (Blood and lymphatic system disorders) | 8 | 30
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 3
Drug hypersensitivity (Immune system disorders) | 1 | 3
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Spinal cord compression (Nervous system disorders) | 8 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 3
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Convulsion (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Corneal erosion (Eye disorders) | 0 | 1
Pigmentary glaucoma (Eye disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 7
Palpitations (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 5 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 5
Hypotension (Vascular disorders) | 3 | 4
Deep vein thrombosis (Vascular disorders) | 6 | 4
Phlebitis superficial (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 2
Hypertensive crisis (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 13
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 17
Stomatitis (Gastrointestinal disorders) | 1 | 14
Nausea (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 5
Haematochezia (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 7
Anal inflammation (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 5
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Ileus (Gastrointestinal disorders) | 0 | 2
Rectal ulcer (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 2
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 3
Peptic ulcer (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Faecalith (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal tract mucosal discolouration (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Mallory-weiss syndrome (Gastrointestinal disorders) | 0 | 1
Necrotising colitis (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Omental infarction (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Periproctitis (Gastrointestinal disorders) | 1 | 0
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 0 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 5
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Ureteric haemorrhage (Renal and urinary disorders) | 0 | 1
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 0 | 5
Asthenia (General disorders) | 3 | 6
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 6 | 8
Pain (General disorders) | 0 | 1
Disease progression (General disorders) | 3 | 10
Non-cardiac chest pain (General disorders) | 1 | 1
Infusion site extravasation (General disorders) | 0 | 1
Performance status decreased (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Death (General disorders) | 1 | 2
Injection site reaction (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 1
Sudden death (General disorders) | 0 | 2
Sudden cardiac death (General disorders) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Electrocardiogram t wave inversion (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Electrocardiogram st-t segment abnormal (Investigations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 2
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Urinary bladder rupture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=598) | Aflibercept (N=611)
Urinary tract infection (Infections and infestations) | 38 | 39
Nasopharyngitis (Infections and infestations) | 36 | 23
Decreased appetite (Metabolism and nutrition disorders) | 110 | 190
Insomnia (Psychiatric disorders) | 44 | 45
Dysgeusia (Nervous system disorders) | 107 | 108
Headache (Nervous system disorders) | 45 | 95
Neuropathy peripheral (Nervous system disorders) | 76 | 56
Peripheral sensory neuropathy (Nervous system disorders) | 75 | 51
Paraesthesia (Nervous system disorders) | 49 | 38
Dizziness (Nervous system disorders) | 50 | 29
Lacrimation increased (Eye disorders) | 71 | 119
Hypertension (Vascular disorders) | 66 | 207
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 36 | 230
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 55 | 199
Cough (Respiratory, thoracic and mediastinal disorders) | 77 | 111
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 89
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 69
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 17 | 38
Diarrhoea (Gastrointestinal disorders) | 209 | 268
Stomatitis (Gastrointestinal disorders) | 123 | 340
Nausea (Gastrointestinal disorders) | 166 | 165
Constipation (Gastrointestinal disorders) | 131 | 133
Vomiting (Gastrointestinal disorders) | 84 | 90
Abdominal pain (Gastrointestinal disorders) | 45 | 47
Dyspepsia (Gastrointestinal disorders) | 29 | 31
Haemorrhoids (Gastrointestinal disorders) | 14 | 31
Dysphagia (Gastrointestinal disorders) | 1 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 268 | 224
Nail disorder (Skin and subcutaneous tissue disorders) | 97 | 94
Rash (Skin and subcutaneous tissue disorders) | 33 | 49
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 51
Back pain (Musculoskeletal and connective tissue disorders) | 83 | 55
Arthralgia (Musculoskeletal and connective tissue disorders) | 66 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 62 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 58 | 41
Bone pain (Musculoskeletal and connective tissue disorders) | 44 | 35
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 33 | 21
Muscle spasms (Musculoskeletal and connective tissue disorders) | 31 | 17
Proteinuria (Renal and urinary disorders) | 6 | 31
Fatigue (General disorders) | 241 | 243
Asthenia (General disorders) | 123 | 144
Oedema peripheral (General disorders) | 157 | 57
Pyrexia (General disorders) | 54 | 61
Weight decreased (Investigations) | 51 | 201

LIMITATIONS AND CAVEATS:
Pain response initially defined as a key secondary endpoint together with PSA response, time to occurence of SRE and PFS was finally considered as an exploratory endpoint in final statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission to a journal, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).